CLINICAL TRIAL: NCT06992310
Title: Exploration of the Functional Effect of Different Hearing Aid Noise Reduction Algorithms in an Ecologically Valid Conversational Situation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastian Griepentrog (Industry)
Responsible Party: Sponsor-Investigator, Sebastian Griepentrog, Clinical studies manager, Sonova AG
Organization: Sonova AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-30177
Record Dates: First submitted 2025-05-27; First posted 2025-05-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with each sound changing principle in a randomized order.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hearing aid standard NR_1 (Active Comparator): Hearing Aid with standard noise reduction (NR) serves as reference condition
  Interventions: Device: Hearing Aid with standard noise reduction (NR_1)
- Hearing Aid with NR_2 (Experimental): NR_2: Noise reduction principle 2
  Interventions: Device: Hearing Aid with NR_2
- Hearing Aid with NR_3 (Experimental): NR_3: Noise reduction principle 3
  Interventions: Device: Hearing Aid with NR_3

INTERVENTIONS:
Device: Hearing Aid with standard noise reduction (NR_1) — Each participant will be fitted with the 3 different noise reduction (sound changing) principles on the same hearing aid, saved to 3 manual programs (ensures exact same hearing loss compensation for each intervention).
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort.
  The active comparator condition is the state of the art Noise Reduction principle to mimic the natural directivity of the outer ear.
  Arms: Hearing aid standard NR_1
Device: Hearing Aid with NR_2 — Each participant will be fitted with the 3 different noise reduction (sound changing) principles on the same hearing aid, saved to 3 manual programs (ensures exact same hearing loss compensation for each intervention).
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort.
  The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Arms: Hearing Aid with NR_2
Device: Hearing Aid with NR_3 — Each participant will be fitted with the 3 different noise reduction (sound changing) principles on the same hearing aid, saved to 3 manual programs (ensures exact same hearing loss compensation for each intervention).
  Noise Reduction principle is a sound processing algorithm to remove noise from a speech signal to improve the speech intelligibility and comfort.
  The experimental conditions vary in their parametrization to result in different degrees of noise suppression and good speech quality.
  Arms: Hearing Aid with NR_3

SUMMARY:
A methodical evaluation of sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and asses strength and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Objective laboratory measurements as well as subjective ratings will be carried out. This will be a controlled, single blinded and randomized active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa.

ELIGIBILITY:
Inclusion Criteria:

* Good written and spoken German language skills
* No suffering from any speech disorders
* Experienced hearing aid user (min. 6 months)
* Ability to stand and walk during the experiment
* Ability to fill in a questionnaire conscientiously
* Ability to produce a reliable hearing test result
* Ability to describe listening experiences/impressions
* The audiogram is in the fitting range of the hearing aid
* The audiogram is in the range of mild to moderate hearing losses (N2 - N4)
* Hearing loss in both ears
* Informed consent form

Exclusion Criteria:

* Contraindications to the medical device
* Unaidable hearing loss in one or both ears
* Acute tinnitus (in either one ear and occurrence for less than 3 months)
* Anatomical deformity of one or both ears
* Single-sided deafness
* Unwillingness to wear the investigational device during the investigational visits
* Active pacemaker implant
* Ear canals are too narrow to take ear impressions
* Ear canals are too narrow for the use of customized earpieces
* Uncomfortable loudness threshold less than 80 dB for at least one measured frequency
* Known hypersensitivity or allergy against synthetic materials
* Acute symptoms of vertigo or dizziness
* Reported Parkinson's disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Own Voice Level | 3 weeks
  Changes to the participants' own voice level (RMS in dB) during a conversation in noise in the laboratory will be recorded in each interventional condition.

SECONDARY OUTCOMES:
Interpersonal distance | 3 weeks
  Changes to the participants' interpersonal distance (in m) during a conversation in noise in the laboratory will be measured in each interventional condition.
Qualitative interview form | 3 weeks
  A qualitative questionnaire with predefined questions to gather individual perceptions regarding the 3 interventional conditions during a conversation in noise in the laboratory. The data collected from this questionnaire are scores on a rating scale from "0" (worst) to "5" (best) in increments of 1.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Hollenbach, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No